CLINICAL TRIAL: NCT02859233
Title: Role of Prophylaxis by Oral Fluid Supplementation in Prevention of Postdural Puncture Headache: A Non-inferiority Randomized Controlled Trial
Brief Title: Role of Prophylaxis by Oral Fluid Supplementation in Prevention of Postdural Puncture Headache
Acronym: PROPHYDRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC16_0031
Record Dates: First submitted 2016-07-21; First posted 2016-08-09 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Postdural Puncture Headache
Keywords: Spinal Puncture; Dural puncture; Nursing
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Routine advices about the interest of increase fluid after lumbar puncture to prevent PDPH will be transmitted: 2 liters will be provided to be drunk in 2 hours.
- Interventional group (Experimental): Lack of hyperhydration : no particular advices will be transmitted about the interest of oral hyperhydration. 500 milliliters will be provided in case of thirst, according to patient's convenience.
  Interventions: Other: Lack of hyperhydration

INTERVENTIONS:
Other: Lack of hyperhydration
  Arms: Interventional group

SUMMARY:
Postdural puncture headache (PDPH) is defined, according to the International Headache Society, as any headache develops within 5 days after a lumbar puncture. It worsens within 15 minutes after sitting or standing and improves within 15 minutes after lying.

For preventing PDPH, there are some uncomfortable practices for patients (fluid supplementation and bed rest) and expensive for hospital (time spend for information and management of fluid intake). Patients are usually advised by nurses. If "bed rest" is not effective in prevention of PDPH, "fluid supplementation" is not an advice based on any evidence but only on routine. By this trial, the investigators want to evaluate the scientific value of this advice, in the standard patient care.

The primary objective of this study is to compare oral hyperhydration (2 liters during 2 hours after lumbar puncture - the most common routine according to an internal pilot survey) versus no advice about the fluid intake to prevent the PDPH.

The second objective is to observe the day of apparition of PDPH, between day 0 and day 5.

DETAILED DESCRIPTION:
Postdural puncture headache (PDPH) is defined, according to the International Headache Society, as any headache develops within 5 days after a lumbar puncture. It worsens within 15 minutes after sitting or standing and improves within 15 minutes after lying.

For preventing PDPH, there are some uncomfortable practices for patients (fluid supplementation and bed rest) and expensive for hospital (time spend for information and management of fluid intake). Patients are usually advised by nurses. If "bed rest" is not effective in prevention of PDPH, "fluid supplementation" is not an advice based on any evidence but only on routine. By this trial, the investigators want to evaluate the scientific value of this advice by non-inferiority study, in the standard patient care.

The primary objective of this study is to compare oral hyperhydration (2 liters during 2 hours after lumbar puncture - the most common routine according to an internal pilot survey) versus no advice about the fluid intake to prevent the PDPH. It will be evaluated on the occurrence of PDPH in both of the two groups The second objective is to observe the day of apparition of PDPH, between day 0 and day 5.

ELIGIBILITY:
Inclusion Criteria:

* Patient in need of dural puncture for diagnostic.
* Age between 18 and 60 years old.
* Patient willing to participate in the research.

Exclusion Criteria:

* Pregnancy.
* Contraindication for increased oral fluid intake.
* Previous dural puncture within 5 day prior enrollment.
* Parenteral fluid intake superior at 266 ml for 2 hours after dural puncture (1000 ml per day).
* Enteral artificial feeding.
* Patient not in capacity to understand correctly French.
* Patient whose cannot be followed correctly by phone.
* Patient refusing to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
The incidence of PDPH. | At D5
  PDPH will be observed on the 5th day (D5) after the lumbar puncture (D0). If PDPH is still present on the 5th day, the patient continues to be followed until the 8th day after the lumbar puncture
The incidence of PDPH (in case of PDPH still present at D5). | At D8
  PDPH will be observed also on the 8th day (D8) after the lumbar puncture (D0). , if PDPH was still present on the 5th day, to confirm the diagnosis of PDPH.

SECONDARY OUTCOMES:
The date of apparition of PDPH between day 0 and day 5 | between day 0 and day 5

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle CARTRON, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Hospital centre CHD VENDEE, La Roche-sur-Yon
  - Hospital centre LE MANS, Le Mans
  - University Hospital NANTES, Nantes
  - Hospital centre CORNOUAILLE, Quimper

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Arevalo-Rodriguez I, Ciapponi A, Roque i Figuls M, Munoz L, Bonfill Cosp X. Posture and fluids for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2016 Mar 7;3(3):CD009199. doi: 10.1002/14651858.CD009199.pub3. PMID 26950232
- [Background] Armon C, Evans RW; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Addendum to assessment: Prevention of post-lumbar puncture headaches [RETIRED]: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2005 Aug 23;65(4):510-2. doi: 10.1212/01.wnl.0000173034.96211.1b. PMID 16116106
- [Background] Dieterich M, Brandt T. Incidence of post-lumbar puncture headache is independent of daily fluid intake. Eur Arch Psychiatry Neurol Sci. 1988;237(4):194-6. doi: 10.1007/BF00449906. PMID 3203698
- [Derived] Cartron E, Volteau C, Leroy M, Voisine A, Dauvergne JE, Ballet C, Talarmin JP, Queau MA, Catinault M, Gazeau E, Haubertin C, Charreau R, Boutoille D. Oral fluid supplementation for the prevention of post-dural puncture headache: A noninferiority randomized controlled trial. PLoS One. 2025 Mar 12;20(3):e0319481. doi: 10.1371/journal.pone.0319481. eCollection 2025. PMID 40073366